CLINICAL TRIAL: NCT05977270
Title: Evaluation of the Effects of Lifebloom One on Physical Activity After Acquired Brain Injury: A Single-Case Experimental Study
Brief Title: The Effects of Lifebloom One on Physical Activity After Acquired Brain Injury
Acronym: LBO_LCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifebloom (Industry)
Collaborators: Pitié-Salpêtrière Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A00072-39
Record Dates: First submitted 2023-07-13; First posted 2023-08-04 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Brain Injuries, Traumatic
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design with multiple baselines across individuals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifebloom One intervention (Experimental)
  Interventions: Device: Lifebloom One

INTERVENTIONS:
Device: Lifebloom One — LBO is made of Oxilio, an alternative to wheelchair placement for everyday use.

SUMMARY:
The goal of this clinical trial is to evaluate the effects of Lifebloom One in people who have suffered a stroke or a traumatic brain injury.

The main questions to be answered are:

* Does Lifebloom One allow users to spend more time standing each day?
* Does Lifebloom One allow users to improve their balance and gait?

Participants will use Lifebloom One during 8 weeks.

For each participant, gait and balance are compared either with and without Oxilio or before and after Lifebloom One intervention.

ELIGIBILITY:
Inclusion Criteria:

* Stroke or traumatic brain injury more than 2 months old
* Unable to walk without assistance
* Expected length of stay equal to or greater than 4 months

Exclusion Criteria:

* Anthropometric incompatibility with Oxilio
* Unable to walk prior to brain injury
* No functional upper limb
* Complete sensory deficit in the lower limb(s)
* Degenerative impairment (tumor, neurodegenerative disease, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Assessment of daily time spent standing change | Change from baseline to intervention phase

SECONDARY OUTCOMES:
10 meter walk test change | Change from baseline to intervention phase
Functional Ambulation Categories (FAC) change | Change from baseline to intervention phase
  6-point scale. A score of 0 indicates that the patient is a non-functional ambulator, a score of 1, 2 or 3 denotes a dependent ambulator who requires assistance from another person in the form of continuous manual contact (1), continuous or intermittent manual contact (2), or verbal supervision/guarding (3) and a score of 4 or 5 describes an independent ambulator who can walk freely on: level surfaces only (4) or any surface (5=maximum score).
Berg Balance Scale change | Change from baseline to intervention phase
  In this 14-item scale, patients must maintain positions and complete moving tasks of varying difficulty. In most items, patients must maintain a given position for a specified time. Patients receive a score from 0-4 on their ability to meet these balance dimensions. A global score can be calculated out of 56. A score of 0 represents an inability to complete the item, and a score of 56 represents the ability to independently complete the item.
Fatigue Severity Scale change | Change from baseline to intervention phase
  A 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity according to a self-report scale. The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
6 minutes walk test | From the beginning and until the end of the intervention phase (during 8 weeks, one time per week)
Barthel Index (BI) | Before baseline, twice during the intervention phase, at immediate post-intervention
  The score of the BI is a summed aggregate and there is preferential weighting on mobility and continence. The scores are allotted in the following way: 0 or 5 points per item for bathing and grooming; 0, 5, or 10 points per item for feeding, dressing, bowel control, bladder control, toilet use, and stairs; 0, 5, 10, or 15 points per item for transfers and mobility. The Index yields a total score out of 100 - the higher the score, the greater the degree of functional independence.
Stroke Specific Quality of Life Scale | Before baseline, at immediate post-intervention
  It is a self-report scale containing 49 items. Items are rated on a 5-point Likert scale. Higher scores indicate better functioning.
Patient Health Questionnaire - 9 | Before baseline, at immediate post-intervention
  The PHQ-9 contains the 9 items. Each item is evaluated on a severity scale ranging from 0 to 3 where the respondent is asked to rate how often each symptom occurred over the last 2 weeks (0-not at all; 1-several days; 2-more than half of the days or 3-nearly every day), yielding a total score ranging from 0-27. Score interpretation:1-4 minimal depression; 5-9 mild depression; 10-14 moderate depression; 15-19 moderately severe depression; and 20-27 severe depression.
Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) | at immediate post-intervention
Psychosocial Impact of Assistive Device Scale (F-PIADS) | at immediate post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Eleonore Bayen, PUPH, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Physical Medicine and Rehabilitation Department - Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No